CLINICAL TRIAL: NCT00003543
Title: Phase I Study of Combination Immunochemotherapy in Patients With Advanced Colorectal Carcinoma
Brief Title: Monoclonal Antibody Therapy Plus Combination Chemotherapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-056; CDR0000066597 (Registry Identifier: PDQ (Physician Data Query)); NCI-H98-0022
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Carmustine; Fluorouracil; Streptozocin; Vincristine

INTERVENTIONS:
Biological: monoclonal antibody A33
Drug: carmustine
Drug: fluorouracil
Drug: streptozocin
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies can find and locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy plus combination chemotherapy in treating patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define toxicity and the maximum tolerated dose of humanized monoclonal antibody A33 (MOAB A33) when combined with carmustine, fluorouracil, vincristine, and streptozocin in patients with advanced colorectal cancer. II. Determine the effect of chemotherapy on human antihuman antibody response and on the pharmacokinetics of humanized MOAB A33 in these patients. III. Define the humanized MOAB A33 dose for a phase II study.

OUTLINE: This is a dose escalation study of humanized monoclonal antibody A33 (MOAB A33). Patients receive humanized MOAB A33 IV once a week for 14 weeks. Chemotherapy begins on day 29 and consists of carmustine IV on days 29-33, fluorouracil IV on days 29-33 and 64-68, vincristine IV on days 29 and 64, and streptozocin IV every 7 days, beginning on day 29, for 10 doses. Courses repeat every 14 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of humanized MOAB A33. The maximum tolerated dose is defined as the dose at which no more than 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: There will be 3-18 patients accrued into this study over 2-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable stage IV colon or rectal cancer that has failed conventional chemotherapy for advanced disease or refused other treatment Measurable disease No liver involvement of greater than 50% No clinical evidence of CNS tumor involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Life expectancy: At least 14 weeks Hematopoietic: WBC at least 3,5000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.0 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No clinically significant cardiac disease (New York Heart Association class III/IV heart disease) Other: No positive human antimouse antibody titer No serious infection requiring treatment with antibiotics No other serious illness Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior mouse monoclonal antibody or antibody fragment, or chimeric or humanized antibody At least 4 weeks since prior immunotherapy Chemotherapy: No prior carmustine, fluorouracil, vincristine, and streptozocin At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Welt, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States